CLINICAL TRIAL: NCT01534806
Title: A Randomized Double Blinded Study Comparing Use of Prochlorperazine Versus Prochlorperazine and Ketorolac in the Treatment of Pediatric Migraine in the Emergency Department
Brief Title: Prochlorperazine Versus Prochlorperazine & Ketorolac in Treatment of Pediatric Migraine in the Emergency Department
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Drug is backordered;
Sponsor: Akron Children's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 110808
Record Dates: First submitted 2011-11-08; First posted 2012-02-17 (Estimated); Last update posted 2014-06-24 (Estimated); Status verified 2014-06

CONDITIONS: Migraine
Keywords: Migraine
MeSH Terms: conditions — Migraine Disorders | interventions — Ketorolac

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ketorolac (Experimental)
  Interventions: Drug: Ketorolac
- Placebo (Placebo Comparator): Placebo IV push
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ketorolac — Ketorolac(0.5mg/kg) IV push
  Arms: ketorolac
Drug: Placebo — Sodium Chloride 0.9% - 10 mL IV push
  Arms: Placebo

SUMMARY:
The aim of this study is to evaluate whether the use of prochlorperazine and ketorolac in combination lead in a larger reduction in pain score compared to prochlorperazine alone when treating pediatric migraine in the Emergency Department (ED). Our hypothesis is that this combination of medications treats not only the pain but also the associated gastrointestinal symptoms of migraine. The main outcome of this study is the reduction in the patient's pain score at 60 minutes from administration of the study medications. Secondary outcomes include the number of patients achieving complete resolution of the headache while in the ED, the number of patients requiring additional treatment interventions by the treating physician, the number of patients with resolution of the associated symptoms like nausea, vomiting, photophobia and phonophobia, the recurrence of headache in the 48-72 hours after discharge, and side effects of the medications.

ELIGIBILITY:
Inclusion Criteria:

1. patient aged 8-18 years presenting to Akron Children's Hospital (ACH) ED with complaint of headache
2. patient has an established diagnosis of migraine without aura or as established by history meets the criteria for migraine headache as defined by the International Criteria for Headache Disorder -II in 2004 a. At least 5 episodes of headache b. The headache should last between 1-72 hours c. The headache should include two of the following: i. Unilateral location, though may be bifrontal or frontotemporal in location but should not be occipital ii. Pulsing quality iii. Moderate to severe pain iv. Aggravation by or causing avoidance of routine physical activity d. One of the following symptoms should accompany the headache i. Nausea or vomiting ii. Photophobia or phonophobia e. The headache should not be attributed to another disorder based on history, physical and/or laboratory information.

Exclusion Criteria:

1. Patients with a contraindication to receiving prochlorperazine, ketorolac, diphenhydramine, or naproxen
2. Patients unable to complete the pain scale.
3. Patients on medications that will have a drug-drug interaction with the study medication including prochlorperazine, ketorolac, diphenhydramine or naproxen.
4. Patients with any medical condition that may be contributing or associated with the current headache such as concussion or trauma
5. Female patients with a positive urine HCG point of care test
6. Patients with diagnosis of or suspected to have chronic daily headaches defined as a headache lasting at least 4 hours for more than 15 days a month for the past 3 months.
7. Patients who received prochlorperazine or ketorolac in the past 48 hours.
8. Patients who had previously been randomized in this study in the past 3 months.

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2012-01; Primary Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Reduction in the patient's pain score at 60 minutes from administration of the study medications | 60 minutes from administration of the study medications

SECONDARY OUTCOMES:
number of patients achieving complete resolution of the headache while in the emergency department. | while in the emergency department, an expected average of 2 hours.
number of patients requiring additional treatment interventions by the treating physician | while in the emergency department, an expected average of 2 hours.
number of patients with resolution of the associated symptoms like nausea, vomiting, photophobia and phonophobia | while in the emergency department, an expected average of 2 hours.
recurrence of headache | 48-72 hours after discharge
side effects of medications | 48-72 hours after discharge

CONTACTS AND LOCATIONS:
Overall Officials: sarah Kline-Krammes, MD, Principal Investigator — Akron Children's Hospital
Locations (1):
- Akron Children's Hospital, Akron, Ohio, United States

REFERENCES:
- [Background] Kan L, Nagelberg J, Maytal J. Headaches in a pediatric emergency department: etiology, imaging, and treatment. Headache. 2000 Jan;40(1):25-9. doi: 10.1046/j.1526-4610.2000.00004.x. PMID 10759899
- [Background] Lewis DW, Qureshi F. Acute headache in children and adolescents presenting to the emergency department. Headache. 2000 Mar;40(3):200-3. doi: 10.1046/j.1526-4610.2000.00029.x. PMID 10759922
- [Background] Lipton RB, Stewart WF, Diamond S, Diamond ML, Reed M. Prevalence and burden of migraine in the United States: data from the American Migraine Study II. Headache. 2001 Jul-Aug;41(7):646-57. doi: 10.1046/j.1526-4610.2001.041007646.x. PMID 11554952
- [Background] Lewis DW. Toward the definition of childhood migraine. Curr Opin Pediatr. 2004 Dec;16(6):628-36. doi: 10.1097/01.mop.0000143763.17125.03. PMID 15548924
- [Background] Hamalainen ML, Hoppu K, Valkeila E, Santavuori P. Ibuprofen or acetaminophen for the acute treatment of migraine in children: a double-blind, randomized, placebo-controlled, crossover study. Neurology. 1997 Jan;48(1):103-7. doi: 10.1212/wnl.48.1.103. PMID 9008503
- [Background] Jones J, Sklar D, Dougherty J, White W. Randomized double-blind trial of intravenous prochlorperazine for the treatment of acute headache. JAMA. 1989 Feb 24;261(8):1174-6. PMID 2915441
- [Background] Coppola M, Yealy DM, Leibold RA. Randomized, placebo-controlled evaluation of prochlorperazine versus metoclopramide for emergency department treatment of migraine headache. Ann Emerg Med. 1995 Nov;26(5):541-6. doi: 10.1016/s0196-0644(95)70001-3. PMID 7486359
- [Background] Seim MB, March JA, Dunn KA. Intravenous ketorolac vs intravenous prochlorperazine for the treatment of migraine headaches. Acad Emerg Med. 1998 Jun;5(6):573-6. doi: 10.1111/j.1553-2712.1998.tb02463.x. PMID 9660282
- [Background] Kabbouche MA, Vockell AL, LeCates SL, Powers SW, Hershey AD. Tolerability and effectiveness of prochlorperazine for intractable migraine in children. Pediatrics. 2001 Apr;107(4):E62. doi: 10.1542/peds.107.4.e62. PMID 11335783
- [Background] Brousseau DC, Duffy SJ, Anderson AC, Linakis JG. Treatment of pediatric migraine headaches: a randomized, double-blind trial of prochlorperazine versus ketorolac. Ann Emerg Med. 2004 Feb;43(2):256-62. doi: 10.1016/s0196-0644(03)00716-9. PMID 14747817
- [Background] Trottier ED, Bailey B, Dauphin-Pierre S, Gravel J. Clinical outcomes of children treated with intravenous prochlorperazine for migraine in a pediatric emergency department. J Emerg Med. 2010 Aug;39(2):166-73. doi: 10.1016/j.jemermed.2008.08.012. Epub 2009 Jan 15. PMID 19150192
- [Background] Trottier ED, Bailey B, Lucas N, Lortie A. Prochlorperazine in children with migraine: a look at its effectiveness and rate of akathisia. Am J Emerg Med. 2012 Mar;30(3):456-63. doi: 10.1016/j.ajem.2010.12.020. Epub 2011 Feb 5. PMID 21296523
- [Background] McGrath PA. The multidimensional assessment and management of recurrent pain syndromes in children. Behav Res Ther. 1987;25(4):251-62. doi: 10.1016/0005-7967(87)90003-9. No abstract available. PMID 3662987
- [Background] Chambers CT, Giesbrecht K, Craig KD, Bennett SM, Huntsman E. A comparison of faces scales for the measurement of pediatric pain: children's and parents' ratings. Pain. 1999 Oct;83(1):25-35. doi: 10.1016/s0304-3959(99)00086-x. PMID 10506669